CLINICAL TRIAL: NCT02510066
Title: Efficacy and Mechanisms of Acupuncture for Patients With Advanced Pancreatic Cancer Pain: : a Randomized, Placebo Controlled Trial
Brief Title: Efficacy and Mechanisms of Acupuncture for Patients With Advanced Pancreatic Cancer Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12401905600
Record Dates: First submitted 2015-07-23; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Pancreatic Cancer; Pain
Keywords: Pancreatic Cancer; Pain; Acupuncture
MeSH Terms: conditions — Pancreatic Neoplasms; Pain | interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Acupuncture participants would receive electroacupuncture on Jiaji (Ex-B2) points for 3 times in a week.
  Interventions: Device: Acupuncture
- Placebo acupuncture (Placebo Comparator): Placebo acupuncture participants would receive placebo acupuncture on non-point points for the same period.
  Interventions: Device: Placebo acupuncture

INTERVENTIONS:
Device: Acupuncture — Disposable stainless steel filiform needles (40mm in length and 0.30mm in diameter) are inserted perpendicularly into T8-T12 Jiaji (Ex-B2) points bilaterally to a depth of 25 mm. After De Qi sensation is achieved, the handles of needles on homolateral T8 and T12 Jiaji are respectively connected to the Han's acupoint nerve stimulator at a frequency of 2/100 Hz and a current of 1mA with a disperse-dense waveform for 30 minutes.
  Other Names: Electroacupuncture
  Arms: Acupuncture
Device: Placebo acupuncture — Placebo acupuncture needles (Dongbang AcuPrime Acupuncture Inc., South Korea) are used on the non-point points at the same level as T8 and T12 Jiaji, 4.5 cun lateral to the posterior median line. The needles with blunt tips are quickly put onto points without inserting into the skin. The needles on homolateral points at the same level as T8 and T12 Jiaji are then connected to the electric stimulator, but with zero frequency and electric current.
  Arms: Placebo acupuncture

SUMMARY:
This study compares the effect of acupuncture and placebo acupuncture on advanced pancreatic cancer pain and then investigates its potential mechanism of peripheral blood.

DETAILED DESCRIPTION:
Acupuncture may alleviate abdominal or back pain of patients with advanced pancreatic cancer. Acupuncture participants would receive electroacupuncture on Jiaji (Ex-B2) points for 3 times in a week. Placebo acupuncture participants would receive placebo acupuncture on non-point points for the same period. Pain scores on numeric rating scale (NRS) and blood levels of β-endorphin and nerve growth factor are compared.

ELIGIBILITY:
Inclusion Criteria:

* Advanced pancreatic cancer at Ⅲ-Ⅳ stage diagnosed by histological/cytological examination.
* Pain score of abdominal or back pain ≥3 on a numeric rating scale (NRS) graduated from 0 to 10.
* Stable dose of analgesics at least 72 hours before randomization.
* Expected survival time more than 1 month.

Exclusion Criteria:

* Another cause for abdominal or back pain (such as prolapse of lumbar intervertebral disc, ulcer or other intra-abdominal disorder).
* Acupuncture treatment in the past.
* Contraindications for the use of acupuncture (such as severe allergies, bleeding tendency, infectious dermatosis and ulcer or scar at points).
* Unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Pain scores, assessed with numeric rating scale (NRS) | 1 week

SECONDARY OUTCOMES:
Karnofsky performance status (KPS) score | 1 week
Blood levels of β-endorphin | 1 week
Blood levels of nerve growth factor | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Hao Chen, Study Chair — Shanghai Cancer Hospital
Locations (1):
- Shanghai Cancer Hospital, Shanghai, Shanghai Municipality, China